CLINICAL TRIAL: NCT06170424
Title: A Real-world 10-year Single Center Experience With Spray Skin in the Treatment of Extensive Severe Burns
Brief Title: Retrospective Analysis of Spray Skin Treats for Severe Burns
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Zhu Jiayuan, Professor, First Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: SYSU-FAH-2019287
Record Dates: First submitted 2023-12-03; First posted 2023-12-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Morality; Skin Graft Complications
Keywords: spray skin, severe burn, microskin grafting
MeSH Terms: conditions — Burns | interventions — Control Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- experimental gourp: The patients who used the autologous skin cell suspension combined with skin grafting.
  Interventions: Procedure: spray skin
- Control group: The patients who used split-thickness skin grafting.
  Interventions: Procedure: Control group

INTERVENTIONS:
Procedure: spray skin — The patients who used the autologous skin cell suspension combined with skin grafting.
  Groups: experimental gourp
Procedure: Control group — The patients who used skin grafting.
  Groups: Control group

SUMMARY:
This study investigated the efficacy of novel approach spray skin for extensive severe burns treatment.

DETAILED DESCRIPTION:
Burns are a global public health problem. This study investigated the efficacy of novel approach spray skin (autologous skin cell suspension combined with split-thickness skin grafting, STSG) for extensive severe burns treatment.

We performed a real-world retrospective analysis of extensive burns patients (> 50% TBSA) from our hospital last 10 years.

ELIGIBILITY:
Inclusion Criteria:

* patients with > 50% TBSA

Exclusion Criteria:

* died within 1 week after admission
* admitted to hospital more than 1 week after injury

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: severe burns patients with > 50% TBSA
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
survival rate | through study completion, an average of 1 year
  Patient survival during hospitalization

SECONDARY OUTCOMES:
complication of skin graft | the take rate in the postoperative day 30, 60, 90
  the survival of grafting skin
length of hospital | through study completion, usually no more than 6 months
  The time during which the patient was hospitalized

CONTACTS AND LOCATIONS:
Overall Officials: Jiayuan Zhu, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- Department of Burn Surgery, The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
Subjects' private information needs to be protected, and contact the investigator if necessary.